CLINICAL TRIAL: NCT07073105
Title: Ultrasonography for Confirmation of Endotracheal Tube Placement in Preterm in Neonatal Intensive Care Unit: Expert Versus Trainee
Brief Title: Tracheal Ultrasound for Confirmation of ETT Placement in NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, Assistant Professor of paediatrics and neonatology , Ain shams University, Ain Shams University
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Tracheal Ultrasound NICU
Record Dates: First submitted 2025-07-06; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Preterm Neonates; Mechanical Ventilation; Endotracheal Tube
Keywords: tracheal ultrasound in preterm neonates for ETT confirmation
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- confirmation of ETT by CXR (Active Comparator): confirmation of ETT site by CXR the gold standard
  Interventions: Diagnostic Test: Chest x-ray
- ETT site confirmation by trainee tracheal ultrasound (Experimental): confirmation of ETT site was done by tracheal ultrasound performed by a trainee neonatologist after receiving training for the procedure
  Interventions: Diagnostic Test: tracheal ultrasound by trainee neonatologist
- ETT site confirmation by expert tracheal ultrasound (Experimental): confirmation of ETT tube site by expert radiologist performing tracheal ultrasound
  Interventions: Diagnostic Test: tracheal ultrasound ( expert radiologist)

INTERVENTIONS:
Diagnostic Test: tracheal ultrasound ( expert radiologist) — tracheal ultrasound, performed by expert radiologist, for preterm neonates for confirmation of ETT site
  Arms: ETT site confirmation by expert tracheal ultrasound
Diagnostic Test: tracheal ultrasound by trainee neonatologist — tracheal ultrasound, performed by trainee neonatologist ( after receiving training for the procedure) , for preterm neonates for confirmation of ETT site
  Arms: ETT site confirmation by trainee tracheal ultrasound
Diagnostic Test: Chest x-ray — chest xray done for confirmation of ETT site
  Arms: confirmation of ETT by CXR

SUMMARY:
Improper placement of the endotracheal tube during intubation can lead to dangerous complications. It has been reported that chest radiography is the gold standard method for validation of endotracheal tube (ET) position .

This study will compare the effectiveness of endotracheal tube position obtained by ultrasonography vs that obtained by chest X-ray with two operators an expert and a trainee in preterm neonates.

This study will work to the extent that the trainee has the ability to do sonar for premature babies with the same efficiency as an ultrasound specialist.

DETAILED DESCRIPTION:
neonate in the neonatal intensive care unit (NICU) are intubated for different reasons and most of these patients undergo chest X-rays (CXRs) several times during their ICU admission to confirm endotracheal tube (ETT) placement, monitor severity of cardiopulmonary illness, and detect complications of other indwelling devices Although the amount of radiation exposure is minimal with CXRs, exposure to multiple CXRs in NICU patients, especially in preterm, results in accumulated radiation burden over time. This can lead to tissue damage and is associated with an increased risk of malignancy Tracheal ultrasonography is technique for confirmation of proper endotracheal intubation. Potential advantages include detection of both main stem and esophageal intubation and less time to image availability than CXR and less radiation Point of care ultrasound (POCUS) of the anterior neck is increasingly used by emergency physicians and anesthesiologists to detect endotracheal and esophageal intubation. It is more accurate and faster than physical examination and capnography, with adult meta-analyses reporting that it has sensitivities of 93-98%, specificities of 97-98% We will explore effectiveness and reproducibility of tracheal ultrasonography done by in hospital neonatologist trainee in the technique vs the expert radiologist in determination of ET position.

ELIGIBILITY:
Inclusion Criteria:

* Less than 35weeks gestational age
* Invasive mechanical ventilation via ETT.

Exclusion Criteria:

* Upper air way anomalies.
* eligible patients whose care team deemed enrollment will disrupt patient care.

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
time in minutes to receive tracheal ultrasound by trainee neonatologist results for ETT site | 24 hours
  Time taken from giving order to perform the tracheal ultrasound by trainee neonatologist to receiving the results of the imaging
time in minutes to receive CXR results for ETT site | 24 hours
  Time taken from giving order to perform chest x ray to receiving the results of the imaging
time in minutes to receive tracheal ultrasound by expert radiologist results for ETT site | 24 hours
  Time taken from giving order to perform the tracheal ultrasound by expert radiologist to receiving the results of the imaging
reproducibility of results between CXR , expert and trainee tracheal ultrasound | 24 hours
  Accuracy of the findings of the tracheal ultrasound by expert, trainee and chest x ray for the same patient

CONTACTS AND LOCATIONS:
Overall Officials: mariam ibrahim, MD, PHD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
individual participant data can be shared after publication from the corresponding author upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: after publication
Access Criteria: from the coresponding author

REFERENCES:
- [Derived] Ibrahim MJA, Elbarbary MNED, Yacoub GEE, Abdo MAM. Confirmation and reproducibility of endotracheal tube position by tracheal ultrasonography in preterms: expert versus trainee. Eur J Pediatr. 2025 Dec 9;185(1):2. doi: 10.1007/s00431-025-06626-3. PMID 41364152